CLINICAL TRIAL: NCT01619592
Title: The Belgian Quality of Life and Costs Study on Web-based Education for Diabetes Patients on Adaptable Insulin Schedules
Brief Title: Web-based Education for Diabetes Patients on Adaptable Insulin Schedules
Acronym: Telediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Nikolaas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012/321
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes
Keywords: patients; adaptable; insulin; schemes
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): webbased education (telemonitoring)
  Interventions: Device: webbased education (telemonitoring)
- control group (No Intervention): standard care

INTERVENTIONS:
Device: webbased education (telemonitoring) — Patients will be able to transmit their blood glucose values via the Internet to the diabetes professional and they will receive timely feedback. "Timely" will be defined as 'as agreed between the patient and the diabetes professional', e.g. every week on Friday afternoon.
  Arms: Intervention group

SUMMARY:
Inclusion criteria: adult diabetes patients on multiple daily insulin injections or using an insulin pump; Internet users Exclusion criteria: having a severe mental illness Patients will be recruited during the conventional consult. If they want to participate, they will get detailed information regarding the study; after giving consent; they will sign the informed consent form and they will get a unique study number.

The patient will than complete a questionnaire on a secured website (https://) using the unique study number. After completing this questionnaire, the patient will be randomised either into a group 'standard care + direct start with web-based diabetes education' (intervention group) or they will enter into the other group (control) receiving standard care. Three months after the start of the study, all patients will be asked to complete the questionnaire again and the patients into the control group will also get access to 'standard care + web-based diabetes education'. The questionnaire will have to be completed on months 6, year 1 and year 2. At the time of completing the questionnaire, HbA1c will be determined. This is part of the routine examination in each participating hospital (UZGent and AZ Nikolaas). The determination of HbA1c is not study-specific but the value will be taken into the study.

The web-based questionnaire:

Patients will enter on a website including general study-information. They also have to explicitly click a button to proceed to the questionnaire. After clicking on 'I am prepared to participate in the study' they will see a second webpage retrieving some general information. After receiving this real basic information; they will be redirected to a secure website (https://) and will make use of a unique study number. Only the main researcher will have the possibility to link the general information to the unique study number.

The informed consent form:

The patient will be asked for added information. He/she will have to sign specific pages giving explicitly informed consent for information retrieved from the 'mutualiteit' (National Health Service - NHS).

On the NHS information will be asked regarding the health costs. These figures should make it possible to have a more objective figure of the costs associated to diabetes (care).

The patient can stop on every moment the study participation. Once decided he/she wants to stop, he/she will receive standard care.

Study hypotheses: the QoL will improve by the use of web-based diabetes education; there will be a reduction in costs using web-based diabetes education; there will be at least an equal-stay or improvement of the HbA1c while using web-based diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* adult diabetes patients on multiple daily insulin injections or using an insulin pump;
* Internet users

Exclusion Criteria:

* having a severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | Baseline
  QoL will be measured via validated questionnaires: diabetes self-care questionnaire, Problem Areas in Diabetes, Diabetes Treatment and Satisfaction Questionnaire, Fear for Hypoglycaemia Questionnaire
Quality of Life (QoL) | month 3
  QoL will be measured via validated questionnaires: diabetes self-care questionnaire, Problem Areas in Diabetes, Diabetes Treatment and Satisfaction Questionnaire, Fear for Hypoglycaemia Questionnaire
Quality of Life (QoL) | month 6
  QoL will be measured via validated questionnaires: diabetes self-care questionnaire, Problem Areas in Diabetes, Diabetes Treatment and Satisfaction Questionnaire, Fear for Hypoglycaemia Questionnaire
Quality of Life (QoL) | year 1
  QoL will be measured via validated questionnaires: diabetes self-care questionnaire, Problem Areas in Diabetes, Diabetes Treatment and Satisfaction Questionnaire, Fear for Hypoglycaemia Questionnaire
Quality of Life (QoL) | year 2
  QoL will be measured via validated questionnaires: diabetes self-care questionnaire, Problem Areas in Diabetes, Diabetes Treatment and Satisfaction Questionnaire, Fear for Hypoglycaemia Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ruige, MD, Phd, Study Director — University Hospital, Ghent; Heidi Buysse, Phd, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - AZ Nikolaas: Department of Endocrinology, Sint-Niklaas